CLINICAL TRIAL: NCT03707249
Title: Effects of Iron Status, Manipulated Using Intravenous Iron, on Cardiopulmonary Physiology During Ascent to Very High Altitude
Brief Title: Iron Status and Cardiopulmonary Physiology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Centre for Defence Medicine (Other Government)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Lieutenant Colonel David Holdsworth, Lecturer in Military Medicine, Consultant Cardiologist and General Physician, Royal Centre for Defence Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 663/MODREC/15
Record Dates: First submitted 2018-10-01; First posted 2018-10-16 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Iron-deficiency; Ventricular Function; Pulmonary Vascular Resistance Abnormality; Altitude Hypoxia
MeSH Terms: conditions — Anemia, Iron-Deficiency; Altitude Sickness | interventions — ferric carboxymaltose; Saline Solution

STUDY DESIGN:
Intervention Model Description: 2 groups were randomised to receive a dose of intravenous iron or iv saline control to manipulate body iron stores. They were subsequently investigated non-invasively and with venous blood sampling during an ascent to very high altitude.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants were blinded by the use of eye-masks during infusion and the physical covering of infusion bags and giving sets. Investigators were unaware of the allocation to iron or saline control. Outcomes assessors were also unaware of the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron (Experimental): Received a blinded single 15 mg/kg dose of iv ferric carboxymaltose (Ferinject) up to a maximum off 1g total dose 2 weeks prior to ascent to very high-altitude.
  Interventions: Drug: Ferric Carboxymaltose Injectable Product
- Saline control (Sham Comparator): Received a blinded single dose of iv normal saline 2 weeks prior to ascent to very high-altitude.
  Interventions: Drug: Normal Saline 0.9% Infusion Solution Bag

INTERVENTIONS:
Drug: Ferric Carboxymaltose Injectable Product — iv iron infusion: 15 mg / kg up to a maximum 1g dose of Ferinject diluted in normal saline (0.9%) up to a total volume of 250 ml
  Other Names: Ferinject
  Arms: Iron
Drug: Normal Saline 0.9% Infusion Solution Bag — 250 ml of normal (0.9%) saline given by intravenous infusion over 20 minutes. This constitutes the control for the iron infusion.
  Arms: Saline control

SUMMARY:
This study involved human volunteers undertaking a high-altitude expedition. It assessed changes in physiological parameters of relevance to high-altitude cardiopulmonary physiology. Participants included a subgroup of those taking part in an existing adventurous training expedition and were randomised in a 1:1 fashion to receive either intravenous iron or normal saline several weeks prior to departure. During the expedition, participants were investigated by means of transthoracic echocardiography, peripheral oxygen saturation measurement and heart rate monitoring and through the drawing of venous blood samples. Bloods were later analysed for markers of iron status.

DETAILED DESCRIPTION:
Aim

The aim of the study was to investigate the effects of iron status on human cardiopulmonary physiology during ascent to very high altitude. Differences in iron status were brought about using intravenous iron, and outcomes were assessed using echocardiography and self-reported functional performance scores.

Objectives

Principal objective: To compare echocardiographic parameters in individuals of differing iron status during the expedition.

Secondary objectives: To compare physiological variables (oxygen saturation, pulse) and self-reported functional measures, in individuals of differing iron status during the expedition.

Hypotheses

The primary hypothesis was that iron status, manipulated using intravenous iron, would influence the echocardiographic indices of cardiopulmonary physiological function over the course of the ascent.

A secondary hypothesis was that iron status would influence cardiopulmonary responses in terms of pulse and oxygen saturation, and additionally the perceived exertion involved in ascent to very high altitude.

Design of the Study

The study randomised 18 individuals to iron or normal saline in a 1:1 ratio giving two groups of 9 people. The randomised infusion (control or iron) was undertaken at a pre-expedition meeting approximately 2 weeks prior to the flight to Nepal. The profile of ascent to high altitude will followed internationally accepted acclimatisation guidelines.

Preliminary Testing

To exclude elevated iron stores prior to enrollment, participants underwent an initial blood test. At the pre-exercise mounting station, prior to the flight to Nepal, baseline echocardiography was performed, and blood samples were collected immediately prior to randomisation and infusion. All blood samples in the study were analysed for full blood count, ferritin, iron, transferrin and C-reactive protein (CRP).

Expedition-based tests

Waking peripheral oxygen saturation (%) of haemoglobin (SpO2) and pulse were recorded daily. Venous blood samples were taken for later analysis of variables relevant to iron homeostasis including full blood count, erythropoietin, soluble transferrin receptor and hepcidin. These samples were taken in Kathmandu on the morning following arrival, at the intermediate staging camp (~3,200m) and then at the Dhaulagiri base camp on arrival and after descents from 6,000m and 7,000m.

Measures of both left and right heart function were performed and included: pulmonary artery systolic pressure, pulmonary acceleration time, pulmonary regurgitation end diastolic velocity and tricuspid annular plane systolic excursion (distance of systolic excursion of the right ventricular annular plane towards the apex - TAPSE). Echo parameters were acquired and processed by an appropriately experienced researcher. Measures were taken during exercise on arrival at each test altitude and at rest the following morning. Measurements taken from climbers returning from either 6,000 m or 7,000 m were taken as soon as possible after their return to base camp.

Subjective ratings scales include those for breathlessness (Borg 1-10) and perceived exertion (Borg 6-20).

Blood sample storage and analysis

Once drawn, venous blood was placed on ice. Following centrifugation (3,500 rpm for 10 minutes at 4OC), aliquots of plasma were stored in cryogenic vials at -20°C. Samples drawn at high altitude were transported on dry ice or in liquid nitrogen 'dry-shippers' (safe liquid nitrogen containers that cannot leak nitrogen as liquid) back to the UK (United Kingdom). Subsequent analysis was performed at the University of Oxford.

Statistical analysis

Data were analysed using statistical tests with International Business Machines (IBM) 'statistical package for social sciences' (SPSS) version 22 software.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-pregnant adults
* Age 18-55 years
* Serving in the UK Armed Forces
* Selected for a military mountaineering team intending to climb to very high altitude

Exclusion Criteria:

* Diabetes
* Any cardiovascular or respiratory illness
* Regular medication which would interfere with any outcome measures in the study
* Pregnancy
* Any condition which precludes the administration of Ferinject:

  (i) hypersensitivity to the active substance, to Ferinject® or any of its excipients (ii) known serious hypersensitivity to other parenteral iron products (iii) microcytic anaemia not attributable to iron deficiency (e.g. sickle cell anaemia) (iv) evidence of iron overload or disturbances in the utilisation of iron.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Change in right ventricular systolic pressure (RVSP) with altitude | Measurement performed at baseline (2 weeks prior to commencing ascent to very high altitude) and at intervals during ascent to very high altitude (over a period of 2 weeks)
  Non-invasive measurement of Right ventricular systolic pressure (mmHg) estimated from the velocity of tricuspid regurgitation (TR) (m/s) measured during transthoracic echocardiographic (TTE) continuous wave (CW) Doppler assessment of the tricuspid valve regurgitant jet (RVSP = TR velocity^2 * 4)
Change in time from pulmonary valve opening to peak pulmonary flow velocity with altitude | Measurement performed at baseline (2 weeks prior to commencing ascent to very high altitude) and at intervals during ascent to very high altitude (over a period of 2 weeks)
  The time from pulmonary valve opening to peak velocity flow is inversely correlated with pulmonary artery pressure. This time is measured on a pulsed wave (PW) Doppler trace in the parasternal short axis view at the pulmonary valve level. The measurement is a time and the units are ms. Categories are: normal (>130 ms), borderline elevated (100-130 ms), elevated (80-100 ms) and severely elevated (<80 ms).
Change in left ventricular stroke volume (LV SV) with altitude | Measurement performed at baseline (2 weeks prior to commencing ascent to very high altitude) and at intervals during ascent to very high altitude (over a period of 2 weeks)
  The stroke volume of the left ventricle is calculated from 2-D parasternal echocardiographic measurement of the left ventricular outflow tract diameter (LVOT) and pulsed wave (PW) Doppler measurement of the flow through the LVOT during systole. PW of the LVOT allows measurement of the velocity.time integral of the LVOT flow (VTI). This value, when multiplied by the cross sectional area of the LVOT, allows an extimate of stroke volume. SV = (Pi*(radius of LVOT^2))*VTI of LVOT
Change in left ventricular index of myocardial performance (LIMP) with altitude | Measurement performed at baseline (2 weeks prior to commencing ascent to very high altitude) and at intervals during ascent to very high altitude (over a period of 2 weeks)
  This is a non-invasive measurement of left ventricular function made by transthoracic echocardiography (TTE). Tissue Doppler imaging (TDI) is used to measure the behaviour of the left ventricle throughout the cardiac cycle (both systole and diastole). This allows the time (ms) of isovolumic contraction time (ICT), isovolumic relaxation time (IVRT) and ejection time (ET). The LIMP (also known as Tei index) = IVCT+IVRT/ET. It is a global measure of systolic and diastolic function of the heart.
Change in right ventricular index of myocardial performance (RIMP) with altitude | Measurement performed at baseline (2 weeks prior to commencing ascent to very high altitude) and at intervals during ascent to very high altitude (over a period of 2 weeks)
  This is a non-invasive measurement of right ventricular function made by transthoracic echocardiography (TTE). Tissue Doppler imaging (TDI) is used to measure the behaviour of the left ventricle throughout the cardiac cycle (both systole and diastole). This allows the time (ms) of isovolumic contraction time (ICT), isovolumic relaxation time (IVRT) and ejection time (ET). The RIMP = IVCT+IVRT/ET. It is a global measure of systolic and diastolic function of the heart.
Change in tissue Doppler velocity of the Right Ventricle (RV) and Left Ventricle (LV); units: cm/s, with altitude | Measurement performed at baseline (2 weeks prior to commencing ascent to very high altitude) and at intervals during ascent to very high altitude (over a period of 2 weeks)
  Tissue Doppler imaging (TDI) is performed on the ventricular myocardium 1cm apical to the atrioventricular valve annulus (either the tricuspid valve annulus, for the RV assessment, or the LV septum and LV lateral wall adjacent to the mitral valve for the LV assessment). The parameters are peak systolic velocity (s', cm/s), peak velocity during early diastole (e', cm/s) and peak velocity during atrial systole (a', cm/s).
Change in tricuspid annulus planar systolic excursion (TAPSE) with altitude | Measurement performed at baseline (2 weeks prior to commencing ascent to very high altitude) and at intervals during ascent to very high altitude (over a period of 2 weeks)
  This is a Doppler M-mode measurement of the full range of movement of the tricuspid annulus at the right ventricular (RV) free wall throughout the cardiac cycle. It is measured by placing an M-mode cursor through the connection of the tricuspid annulus to the RV free wall and measuring the basal-apical excursion of the annulus at this point, from end diastole until the most apical point that it reaches in systole. It is a measure of systolic RV function. Its units are cm.
Change in right and left ventricular strain with altitude | Measurement performed at baseline (2 weeks prior to commencing ascent to very high altitude) and at intervals during ascent to very high altitude (over a period of 2 weeks)
  Non-invasive tissue Doppler measurements are acquired on apical 4-chamber, apical 2-chamber and apical 3-chamber images throughout 3 cardiac cycles to allow later analysis to determine the longitudinal strain of the right and left ventricle

SECONDARY OUTCOMES:
Change in peripheral oxygen saturation with altitude | Measurement performed at baseline (2 weeks prior to commencing ascent to very high altitude) and at intervals during ascent to very high altitude (over a period of 2 weeks)
  Peripheral oxygen saturation measured using a non-invasive portable, fingertip pulse oximeter
Change in heart rate with altitude | Measurement performed at baseline (2 weeks prior to commencing ascent to very high altitude) and at intervals during ascent to very high altitude (over a period of 2 weeks)
  Heart rate measured by 3 lead ECG monitor connected to a portable transthoracic echocardiography machine
Change in blood ferritin level (ug/L) with altitude | Measurement performed at baseline (2 weeks prior to commencing ascent to very high altitude) and at intervals during ascent to very high altitude (over a period of 2 weeks)
  Venous blood samples analysed for ferritin
Change in haemoglobin level (g/dL) with altitude | Measurement performed at baseline (2 weeks prior to commencing ascent to very high altitude) and at intervals during ascent to very high altitude (over a period of 2 weeks)
  Venous blood samples analysed for haemoglobin
Change in transferrin saturation (%) with altitude | Measurement performed at baseline (2 weeks prior to commencing ascent to very high altitude) and at intervals during ascent to very high altitude (over a period of 2 weeks)
  Venous blood samples analysed for transferrin and iron to allow the calculation of the transferrin saturation, listed as a percentage
Change in soluble transferrin receptor level (nmol/L) with altitude | Measurement performed at baseline (2 weeks prior to commencing ascent to very high altitude) and at intervals during ascent to very high altitude (over a period of 2 weeks)
  Venous blood samples analysed for soluble transferrin receptor
Change in hepcidin level (ng/mL) with altitude | Measurement performed at baseline (2 weeks prior to commencing ascent to very high altitude) and at intervals during ascent to very high altitude (over a period of 2 weeks)
  Venous blood samples analysed for hepcidin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holdsworth DA, Frise MC, Bakker-Dyos J, Boos C, Dorrington KL, Woods D, Mellor A, Robbins PA. Iron bioavailability and cardiopulmonary function during ascent to very high altitude. Eur Respir J. 2020 Sep 17;56(3):1902285. doi: 10.1183/13993003.02285-2019. Print 2020 Sep. PMID 32430412